CLINICAL TRIAL: NCT06199284
Title: Safety and Efficacy of the Atalante Exoskeleton in the Rehabilitation of Patients With Amyotrophic Lateral Sclerosis: Study Protocol for an Open, Uncontrolled Interventional Study, EXALS.
Brief Title: Atalante Exoskeleton in the Rehabilitation of Patients With Amyotrophic Lateral Sclerosis
Acronym: EXALS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment is suspended due to funding issues
Sponsor: Institut de Recherche sur la Moelle épinière et l'Encéphale (Other)
Collaborators: Association pour la Recherche sur la Sclérose Latérale Amyotrophique et autres Maladies du Motoneurone (Unknown); Groupe Hospitalier Pitie-Salpetriere (Other); Institut de Myologie, France (Other); Station Debout (Unknown); Laboratory of Biomedical Imaging (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A00553-42
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: ALS - Amyotrophic Lateral Sclerosis
Keywords: Atalante exoskeleton; Gait training; Amyotrophic lateral sclerosis; Rehabilitation; Robotics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 3 phases, each lasting 6 weeks, following the ABA procedure. Phase B represents the intervention phase, during which patients will practice their gait training at a rhythm of 3 sessions/week, as an add-on to usual care. In the two phases A, patients receive usual care with no additional treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Other): Single-group study following an ABA design:
  Phase A1 (usual care for 6 weeks) Phase B (usual care + gait training using exoskeleton for 6 weeks) Phase A2 (usual care for 6 weeks) All participants undergo the same sequence of conditions according to the protocol.
  Interventions: Device: Atalante exoskeleton

INTERVENTIONS:
Device: Atalante exoskeleton — The gait training program using Atalante exoskeleton consisted of 3 sessions per week for 6 weeks. Each session includes the patient's installation and de-installation (10 min), walking training (30 min), and physical activities at the end of the session where the patient is in an upright position in the exoskeleton (e.g. badminton, boxing, or basketball) (5-10 min). For each participant, the assistance of the exoskeleton can be specifically adjusted and can be set symmetrically or asymmetrically bases on his capabilities.

SUMMARY:
Using a MRI gait motor imagery paradigm in ALS patients in order to study how ALS affects the function of the central neural networks involved in gait function, we showed a reorganization of the motor networks that represents a compensatory response to the dysfunction of the networks involved in gait function. Our main hypothesis is that by providing coherent proprioceptive input to the sensorimotor integration areas, gait training with an exoskeleton may boost compensatory network reorganization and help to maintain function. We hypothesize that this can be achieved through a locomotion training strategy that reproduces normal gait motor patterns and appropriate sensory feedback. Gait training with an exoskeleton can meet these needs. The Atalante exoskeleton offers unique potential thanks to its cutting-edge technological features, hands-free functions and availability in numerous centers across Europe. Evaluation of its safety and efficacy in ALS is of the utmost interest in order to generalize this new approach in ALS.

DETAILED DESCRIPTION:
Current research is mainly focused on evaluating the effect of robotic rehabilitation on locomotion in ALS. In order to understand this approach, it is important to validate its safety and to determine patient's experience with this new rehabilitation concept in ALS. In this study, we aim to evaluate the safety, the participant experience and effectiveness of the training program with the Atalante exoskeleton as a gait training tool for ALS patients, compared with usual care, on walking ability, functional capacity and other symptoms associated with motor disability. The Atalante exoskeleton is the only self-balancing exoskeleton that enables assisted walking without walking aid, reproducing a natural walking pattern and multidirectional movement. EXALS is an interventional, monocentric, prospective, open trial. With a limited number of studies on gait rehabilitation exoskeletons in ALS, this study represents a significant scientific contribution, being the first to explore the benefits of a self-balancing exoskeleton with a rigorous design. In addition to robust outcome measures, this study places importance on participants' perception, motivation, and involvement in decision-making, adding depth and strength to the research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with amyotrophic lateral sclerosis (defined according to the El Escorial criteria: possible, probable or definite), at the time of diagnosis
* Male or female, between 18 and 70 years of age
* Slowly and moderately evolving patients ∆ ALS Progression rate (FS) ≤ 1.11 (The ALS progression rate was calculated as follows: (48 - ALSFRS-R at screening visit) / (duration from onset to this visit (month)) (Kimura et al., 2006). ALSFRS-R progression will be classified as slow (∆FS ≤ 0.47), intermediate (0.47 ≤ ∆PR ≤1.11) or fast (∆PR > 1.11) (Labra et al., 2016).
* Manual muscle testing ≥ 3 for deltoid muscle and ≥ 4 for neck flexors and extensors muscles
* Ambulatory status: a stable gait deficit with a total score between 3 and 6 on the ALSFRS-R sub-items "walking" and "climbing stairs"
* French speaking patient
* Patient affiliated with the French social security system
* Signed informed consent
* Measurements related to the use of the Atalante exoskeleton:
* Height between 155 and 190 cm
* Weight < 90 kg
* Pelvis width < 46 cm in seated position
* Thigh length between 56.8 and 64.8 cm
* Leg length > 45.7cm or less than:
* 60.7cm if ankle dorsi flexion is ≥16°
* 57.7cm if ankle dorsi flexion is ≥13°and <16°
* 56.7cm if ankle dorsi flexion is>10°and ≤13°
* 55.7cm if ankle dorsi flexion is ≥ 0°and ≤10°
* Joint amplitudes of lower limbs :
* Hip: flexion 90°, extension 5°, medial rotation 10°, lateral rotation 20°, abduction 17°, adduction 10°
* Knee: flexion 5-110°
* Ankle: dorsiflexion (knee straight) 0°, plantarflexion 9°, eversion18°, inversion 18°.

Exclusion Criteria:

* Osteoporosis at the femoral and/or lumbar level (T score ≤ -2.5), confirmed by bone densitometry at both the femoral and lumbar sites.
* Pressure ulcers in areas of contact with the exoskeleton
* Severe spasticity (greater than Ashworth 3) for adductor, hamstring, quadriceps and sural triceps muscles or uncontrolled clonus
* Cardiac or respiratory contraindications to physical effort
* Cognitive impairment that can affect comprehension
* Pregnancy or attempted pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Safety of Atalante exoskeleton | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 and during all training sessions in phase B
  Monitoring adverse events

SECONDARY OUTCOMES:
Functional capacity | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  ALSFRS-R
Pulmonary function | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  Forced vital capacity
Gait ability | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)l
  The 6-minute walk test, the 10-meter walk test and the Timed Up and Go test
Static and dynamic balance | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  Berg Balance Scale (0 - 56) with higher scores representing better balance
Speed of movement of the center of pressure per second | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  Force platform
Lower limb muscle strength | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  Isometric dynamometer
Spasticity of knee flexor and extensor muscles | During the three consecutive phases of the study (A1, B, and A2), from baseline (Week 0) through Week 18, with assessments at Weeks 0, 3, 6, 9, 12, 15, and 18 (7 assessments in total)
  Instrumental assessment with isokinetic dynamometer
Patient quality of life | During the three consecutive phases (A1, B, and A2), with assessments at baseline (Week 0), Week 6, Week 12, and Week 18 (4 assessments in total)
  ALSAQ-40
General fatigue | During the three consecutive phases (A1, B, and A2), with assessments at baseline (Week 0), Weeks 3, 6, 12, and 18 (5 assessments in total).
  Fatigue Severity Scale and the Modified Fatigue Impact Scale
Patient pain | During the three consecutive phases (A1, B, and A2), with assessments at baseline (Week 0), Week 6, Week 12, and Week 18 (4 assessments in total).
  Brief pain inventory-short form
Anxiety and depression | During the three consecutive phases (A1, B, and A2), with assessments at baseline (Week 0), Week 6, Week 12, and Week 18 (4 assessments in total).
  Hospital anxiety and depression scale
Intrinsic motivation | week 12
  Intrinsic motivation inventory
Subjective impact of gait training with Atalante exoskeleton on participants | week 12
  The participant's experience with domain-oriented exoskeleton training
Participants' attitudes to Atalante gait training | week 12
  Net promoter score
Efficacy and interactivity of the Atalante exoskeleton | Week 12
  A specific questionnaire was developed to assess the efficacy and interactivity of the Atalante exoskeleton
Participants' experience of gait training with Atalante exoskeleton | week 12
  Semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Ghida TRAD, PhD, Study Chair — Sorbonne Université, Inserm, CNRS, Laboratoire d'Imagerie Biomédicale (LIB), 75006-Paris (France), Neuromuscular Physiology and Evaluation Lab, Neuromuscular Investigation Center, Institute of Myology, 75013-Paris (France)
Locations (3):
- France (3):
  - Station Debout, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Institut de myologie, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification, may be made available upon reasonable request from the corresponding author. Data sharing will be subject to institutional and ethical approvals.
Supporting Information: Study Protocol
Time Frame: Following publication of the study results
Access Criteria: Researchers with a methodologically sound proposal and appropriate ethical approval may request access to the de-identified data and supporting documents from the corresponding author

REFERENCES:
- [Result] Labra J, Menon P, Byth K, Morrison S, Vucic S. Rate of disease progression: a prognostic biomarker in ALS. J Neurol Neurosurg Psychiatry. 2016 Jun;87(6):628-32. doi: 10.1136/jnnp-2015-310998. Epub 2015 Jul 7. PMID 26152368
- [Result] Kimura F, Fujimura C, Ishida S, Nakajima H, Furutama D, Uehara H, Shinoda K, Sugino M, Hanafusa T. Progression rate of ALSFRS-R at time of diagnosis predicts survival time in ALS. Neurology. 2006 Jan 24;66(2):265-7. doi: 10.1212/01.wnl.0000194316.91908.8a. PMID 16434671
- [Result] Abidi M, de Marco G, Grami F, Termoz N, Couillandre A, Querin G, Bede P, Pradat PF. Neural Correlates of Motor Imagery of Gait in Amyotrophic Lateral Sclerosis. J Magn Reson Imaging. 2021 Jan;53(1):223-233. doi: 10.1002/jmri.27335. Epub 2020 Sep 7. PMID 32896088
- [Derived] Trad G, Lenglet T, Ledoux I, Querin G, Blancho S, Marchand-Pauvert V, Hogrel JY, Pradat PF. Safety and efficacy of the Atalante exoskeleton in the rehabilitation of French patients with amyotrophic lateral sclerosis: a prospective, monocentric, open, uncontrolled, interventional protocol, EXALS. BMJ Open. 2026 Jan 16;16(1):e109620. doi: 10.1136/bmjopen-2025-109620. PMID 41545051